CLINICAL TRIAL: NCT03521648
Title: Database for the Assessment of Efficacy and Safety of BPH Treatment
Acronym: KSSG-BPH-REG
Status: Recruiting | Type: Observational
Sponsor: Dominik Abt (Other)
Responsible Party: Sponsor-Investigator, Dominik Abt, Dr. med. Dominik Abt, Cantonal Hospital of St. Gallen
Organization: Cantonal Hospital of St. Gallen (Other)
Other Study IDs: CTU P-17/006
Record Dates: First submitted 2018-04-29; First posted 2018-05-11 (Actual); Last update posted 2021-01-26 (Actual); Status verified 2021-01

CONDITIONS: Lower Urinary Tract Symptoms; Benign Prostatic Hyperplasia
Keywords: Prostatic Artery Embolization; Transurethral Prostate Resection; Transurethral Electroresection of Prostate; Contact Laser Ablation of Prostate; Laser Enucleation of Prostate; Open prostatectomy
MeSH Terms: conditions — Lower Urinary Tract Symptoms; Prostatic Hyperplasia | interventions — Transurethral Resection of Prostate

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 5 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- PAE: Men with BPH - LUTS BPE who have opted for PAE and have consented to take part in the Register Study.
  Interventions: Procedure: PAE
- TURP: Men with BPH - LUTS BPE who have opted for TURP and have consented to take part in the Register Study.
  Interventions: Procedure: TURP
- Other: Men with BPH - LUTS BPE who have opted for other treatment options (e.g., holmium laser enucleation of the prostate, open prostatectomy, thulium laser vaporization, resection or enucleation, transurethral incision of the prostate) and have consented to take part in the Register Study.
  Interventions: Procedure: Other

INTERVENTIONS:
Procedure: PAE — Prostatic artery embolization
  Groups: PAE
Procedure: TURP — Transurethral resection of the prostate
  Groups: TURP
Procedure: Other — Other surgical procedures for BPH treatment including holmium laser enucleation of the prostate, open prostatectomy, thulium laser vaporization, resection or enucleation, transurethral incision of the prostate
  Groups: Other

SUMMARY:
This registry study aims to collect data on efficacy and safety of different treatments of benign prostatic enlargement (BPE) and lower urinary tract symptoms associated with benign prostatic hyperplasia (BPH-LUTS).

DETAILED DESCRIPTION:
This registry study aims to collect data on efficacy and safety of different treatments of benign prostatic enlargement (BPE) and lower urinary tract symptoms associated with benign prostatic hyperplasia (BPH-LUTS).

Clinical, patient reported and imaging data that are assessed in clinical routine will be prospectively collected. All patients that are treated for BPE / BPH-LUTS at our institution will be included if they provide written informed consent.

This registry enables us to compare novel treatment option (e.g. prostatic artery embolization; PAE) to established interventions (e.g., TURP, HoLEP, open prostatectomy, ThuLEP, Thulium laser vaporization, TUIP) regarding safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

* All patients treated for BPH / LUTS / prostatic obstruction at the urological department of KSSG
* Patient age ≥ 18 years
* Informed consent provided

Exclusion Criteria:

-Cognitive impairment not allowing Informed Consent or adequate data assessment.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All patients treated for BPH / LUTS / prostatic obstruction at the urological department of KSSG
Sampling Method: Probability Sample
Enrollment: 500 (Estimated)
Dates: Start 2017-07-07 (Actual); Primary Completion 2027-12-01 (Estimated); Study Completion 2027-12-01 (Estimated)

PRIMARY OUTCOMES:
Reduction of Lower Urinary Tract Symptoms | baseline to 1 year
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Changes of free urinary flow rate | baseline to 1 year
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of post void residual urine | baseline to 1 year
  Measurement of post void residual urine (mL) by transabdominal ultrasound

SECONDARY OUTCOMES:
Reduction of Lower Urinary Tract Symptoms | baseline to 6 weeks
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | baseline to 12 weeks
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | baseline to 6 months
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | baseline to 2 years
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Reduction of Lower Urinary Tract Symptoms | baseline to 5 years
  Change of total score of International Prostate Symptoms Score (IPSS; range 0 points (no symptoms) to 35 points (severe symptoms))
Changes of free urinary flow rate | baseline to 6 weeks
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | baseline to 12 weeks
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | baseline to 6 months
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | baseline to 2 years
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of free urinary flow rate | baseline to 5 years
  Measurement of urinary stream (mL/s) by urinary flow rate measurement
Changes of post void residual urine | baseline to 6 weeks
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | baseline to 12 weeks
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | baseline to 6 months
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | baseline to 2 years
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Changes of post void residual urine | baseline to 5 years
  Measurement of post void residual urine (mL) by transabdominal ultrasound
Rate of local reinterventions | during 5 year study period
  Assessment of number and type of reinterventions for prostate and bladder problems
Rate of local medical treatment for BPH-LUTS | during 5 year study period
  Assessment of number and type of medical treatments for prostate and bladder problems
Adverse Events | 6 weeks after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 12 weeks after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 6 months after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 1 year after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 2 years after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Adverse Events | 5 years after intervention
  Assessment of adverse events that are at least possibly related to study procedure according to Clavien-Dindo and CTCAE
Urodynamic changes | during 5 year study period
  Results of pressure flow studies if assessed for clinical reasons during the study period
Change of prostate size | 6 weeks after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
Change of prostate size | 12 weeks after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
Change of prostate size | 6 moths after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
Change of prostate size | 1 year after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
Change of prostate size | 2 years after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
Change of prostate size | 5 years after intervention
  Measurement of prostate size (using MRI or ultrasound) in mL
PSA | 6 weeks after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
PSA | 12 weeks after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
PSA | 6 moths after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
PSA | 1 year after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
PSA | 2 years after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
PSA | 5 years after intervention
  Changes of Prostate Specific Antigen (PSA, ng/mL)
Assessment of erectile function | 6 weeks after intervention
  Assessment of IIEF-5 questionnaire
Assessment of erectile function | 12 weeks after intervention
  Assessment of IIEF-5 questionnaire
Assessment of erectile function | 6 moths after intervention
  Assessment of IIEF-5 questionnaire
Assessment of erectile function | 1 year after intervention
  Assessment of IIEF-5 questionnaire
Assessment of erectile function | 2 years after intervention
  Assessment of IIEF-5 questionnaire
Assessment of erectile function | 5 years after intervention
  Assessment of IIEF-5 questionnaire
Reduction of Prostate symptoms | baseline to 6 weeks
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline to 12 weeks
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline to 6 moths
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline to 1 year
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline to 2 years
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Reduction of Prostate symptoms | baseline to 5 years
  Change of CPSI total score (Chronic prostatitis symptoms score; range 0 points (no symptoms) to 43 points (severe symptoms))
Ejaculatory function | 6 weeks after intervention
  Assessment of ejaculatory function according to CTCAE
Ejaculatory function | 12 weeks after intervention
  Assessment of ejaculatory function according to CTCAE
Ejaculatory function | 6 moths after intervention
  Assessment of ejaculatory function according to CTCAE
Ejaculatory function | 1 year after intervention
  Assessment of ejaculatory function according to CTCAE
Ejaculatory function | 2 years after intervention
  Assessment of ejaculatory function according to CTCAE
Ejaculatory function | 5 years after intervention
  Assessment of ejaculatory function according to CTCAE

CONTACTS AND LOCATIONS:
Locations (1):
- St. Gallen Cantonal Hospital, Sankt Gallen, Canton of St. Gallen, Switzerland

IPD SHARING:
Plan to Share IPD: Undecided
Requests for an anonymized, full data set of physician-level data and statistical code will be considered if the proposed use aligns with public good purposes, does not conflict with other requests, or planned use by the trial steering committee and is contingent on approval from the local ethics committee (EKOS). Requests can be addressed to the corresponding author.